CLINICAL TRIAL: NCT05178992
Title: Impact of a Novel Socially Assistive Robotic Architecture on Engaging Older Adults With Mild Cognitive Impairment, Alzheimer's Disease and Related Dementia in Long Term Care Settings
Brief Title: Use of Socially Assistive Robots for Long Term Care Older Adults With Cognitive Impairment and Apathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Nilanjan Sarkar, David K. Wilson Professor of Engineering, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 210386; R01AG062685 (NIH)
Record Dates: First submitted 2021-12-15; First posted 2022-01-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer Disease
Keywords: Apathy; Robotics; Virtual Reality
MeSH Terms: conditions — Alzheimer Disease; Lethargy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either Usual Activity Program or Usual Activity Program + Robot Activity within each long term care facility. At each site, the order of the robot type (humanoid or dog) will be randomized. Each participant will participate in two sessions/week for 8 weeks (4 weeks with humanoid robot, 4 weeks with dog robot).
Who Masked: Outcomes Assessor
Masking Description: Trained research assistants separate from other research personnel will collect outcomes; these research personnel will be blinded to the hypotheses and group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Socially Assistive Robot Activity (Experimental): Participants will attend two sessions per week and interact with the robot. Four weeks with a humanoid robot and four weeks with a dog robot. Participants can continue to join other activities held within the facility.
  Interventions: Behavioral: Socially Assistive Robot Activity
- Usual Activity Program (Active Comparator): Participants will attend at least two sessions per week at activities held within the facility. They will not be exposed to the robot activities.
  Interventions: Behavioral: Socially Assistive Robot Activity

INTERVENTIONS:
Behavioral: Socially Assistive Robot Activity — Participants will attend two weekly sessions with robot activities. Each session will last 30 minutes. Participants will attend robot sessions for 8 weeks.

SUMMARY:
The objective of this study is to demonstrate the impact of a socially assistive robot system on reducing apathy among cognitively impaired older adults residing in long term care facilities. Earlier phases of this project demonstrated the feasibility and acceptability of the robotic system. First, investigators will improve the social robotic interaction architecture through additional software development, enhance its versatility, and make it easy for non-experts to run. Second, 188 participants will be randomized to either usual activity programs at the long term care facility, or the usual activity programs plus the robotic activities. Researchers will examine the effect on apathy and also plan on examining underlying individual and facility factors that influence the impact of the robotic activities.

ELIGIBILITY:
Inclusion Criteria:

* Residing >3 months in long term care facility
* Evidence of mild cognitive impairment (SAGE score 15-16), mild dementia (SAGE score <15, AD8<2, DSRD<19), or moderate dementia (SAGE <15, AD8>1, DSRD 19-36)
* Symptoms of apathy (Score 30+ on AES-C)

Exclusion Criteria:

* Severe cognitive impairment
* Physically unable to participate
* Unable to provide assent
* Uncorrected vision or hearing
* Never spoke English
* Unable to sit comfortably in chair
* Acutely ill, terminally ill or unresponsive
* Unable to be moved to activity location
* Aggressive or combative

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 142 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2026-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Apathy | Baseline to Week 8
  Apathy Evaluation Scale - Clinician (AES-C) will be used to assess changes in composite apathy score from baseline, Week 4, and Week 8. The AES-C is a validated 18-item instrument used to assess cognitive, behavioral, emotional and other symptoms of apathy. Clinicians rate each item based on verbal and nonverbal information provided by the participant. Item scores range from 1 (not at all characteristic) to 4 (a lot characteristic). Total scores range from 18 to 72 where higher derived scores indicate greater apathy.

SECONDARY OUTCOMES:
Change in Trail Making Test (TMT) | Baseline to Week 8
  The TMT is a well established test of executive function and has two forms. TMT-A consists of a series of numbers in circles displayed randomly on a page; the person links the numbers in sequence. TMT-B consists of numbers (1 to 13) and letters (A to L) inside circles randomly placed on a page; the person alternates in connecting ascending numbers with ascending letters. TMT is scored by time in seconds to complete, up to 5 minutes. TMT-A normal time is 29 seconds and deficient score is >78 seconds. TMT-B average score is 75 seconds and deficient score > 273 seconds.
Change in Animal Fluency Test | Baseline to Week 8
  Verbal fluency tests require verbal ability and executive control processes; the Animal Naming test requires naming 15 animals in 1 minute; thus, less than 15 animals named in 1 minute is considered a deficient score.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that are de-identified and have been used in publications.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 12 months after publications

REFERENCES:
- [Derived] Ghosh R, Khan N, Migovich M, Tate JA, Maxwell CA, Newhouse PA, Scharre DW, Tan A, Mion LC, Sarkar N. Engaging Older Adults and Staff in the Co-Design and Evaluation of Socially Assistive Robot and Virtual Reality Activities for Long-Term Care: User-Centered Study. JMIR Aging. 2025 Dec 2;8:e75288. doi: 10.2196/75288. PMID 41330571